CLINICAL TRIAL: NCT00325520
Title: A Neurocognitive Model of Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Klarman Family Foundation (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5984R; K23MH076195-01A2 (NIH)
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2013-07

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anorexia nervosa: Individuals with anorexia nervosa receiving inpatient treatment
- Healthy controls

SUMMARY:
The purpose of this study is to investigate thought processes and neural mechanisms that may contribute to the development of habitual behaviors. The investigators hypothesize that patients with AN will perform differently than people without eating disorders on a series of neuropsychological tasks and will show different neural activation patterns in functional neuroimaging scans.

DETAILED DESCRIPTION:
Patients with Anorexia Nervosa (AN) have extreme difficulty changing their eating behavior, even when they express desire for change. These behaviors seem to override all other potential responses, and can appear perseverative, or habitual. The purpose of this study is to investigate thought processes and neural mechanisms that may contribute to the development of habitual behaviors. The investigators hypothesize that patients with AN will perform differently than people without eating disorders on a series of neuropsychological tasks and will show different neural activation patterns in functional neuroimaging scans.

ELIGIBILITY:
Inclusion:

* DSM-IV-TR™ diagnosis of anorexia nervosa (restricting or binge-purge subtype), current or prior;
* Age 16-45;
* Inpatient on GCRU
* Medically stable.

Exclusion:

* Any other current major Axis I disorder (including current bulimia nervosa), except major depression;
* History of concussion, seizure disorder, or other neurological illness;
* History of learning disability;
* Acute Suicidality

Healthy comparison group:

Inclusion:

* No current or past psychiatric illness;
* Age 16-45
* No history of binge eating or vomiting;
* Normal weight (80%-120% ideal body weight)

Exclusion:

* Significant medical or neurologic illness(concussion, seizure disorder, learning disability, other neurological illness)
* Current psychotropic medication or medications known to impact cognition

Additional Exclusion Criteria for fMRI:

* Significant Claustrophobia
* Pregnancy
* Indwelling metallic object, non-removable metal jewelry, medicinal patch or recent metallic ink tattoo
* For patients, current psychotropic medications (antidepressants for 2 week (prozac and antipsychotics for 4 weeks)
* For patients, any other current Axis I diagnosis

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with Anorexia Nervosa or Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2006-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Neuropsychological functioning | pre- and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Steinglass, MD, Principal Investigator — New York State Psychiatric Institute